CLINICAL TRIAL: NCT04661254
Title: Treg Cell Therapy in Liver and Kidney Transplantation - Preclinical Validation of Batches of Treg Cells Amplified in Vitro
Acronym: PRE-TREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200733; 2020-A01871-38 (Other: ANSM)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplantation; Liver Transplantation
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphapheresis (Other): Blood is drawn from one of the patient's two arms and passes through a separation circuit. After removing the white blood cells, it is reinjected into the other arm.
  Interventions: Other: Lymphapheresis

INTERVENTIONS:
Other: Lymphapheresis — - From the blood product of lymphapheresis: Autologous naïve regulatory CD45RA+CD4+CD25+FoxP3+ T lymphocytes (Tregs) selected and amplified ex vivo; obtained by selection and sorting of CD4+CD25 +CD127lowCD45RA+ cells, derived from lymphapheresis and amplified ex vivo for 10 +/- 1 days, under cGMP condition in the presence of IL2 and Rapamycin

SUMMARY:
Kidney and liver transplantation requires a fine tuning of immune responses in order to achieve long term operational tolerance with immunosuppressants or immune modulators. Numerous experimental findings indicate that CD4+ FOXP3 expressing regulatory T (Treg) cells play a central role in the induction of tolerance to the grafts indicating that the use of Treg cells may be an innovative therapeutic strategy in kidney transplantation that would enable the diminution of immunosuppressive drugs or even their discontinuation, thus decreasing their risk of adverse events.

As human Treg cells represent less than 10% of CD4+ T cells, and because it has been shown in mice that a dose of 2*104 polyclonal Tregs/g was necessary to induce tolerance in animal models of solid organ transplantation, it is mandatory to expand human Treg cells ex vivo, after isolating them from peripheral blood. The investigators previously defined a protocol for Treg cell isolation and expansion in clinical grade conditions (cGMP) that enabled us to obtain the expected number of expanded cells maintaining high levels of FOXP3 (3).

The investigators therefore hypothesize in humans, as it has been already shown in mice, that the infusion of autologous expanded polyclonal Treg cells would lead to the obtaining of operational tolerance in kidney and liver graft in association with classical immunosuppressants and an expectable diminution of those.

To this end, it is necessary to have pre-clinical batches of expanded Treg cells validated by the National Agency for Medicines and Health Products Safety validate (ANSM). The investigators therefore plan to have 4 batches from 2 liver transplant patients and 2 kidney transplant patients validated.

ELIGIBILITY:
Inclusion Criteria:

For liver transplant patients:

* Liver transplantation carried out for 1 to 3 months for alcoholic cirrhosis;
* Normal liver biological test;
* Normal hepatic morphological assessment;

For kidney transplant patients:

* Renal transplantation carried out for 3 to 6 months for any disease requiring renal transplantation;
* Normal renal biological assessment;
* Normal renal morphological assessment;
* DSA <1500 MFI at inclusion

Common criteria:

* Age ≥ 18 years and ≤ 70 years
* GB ≥1500 / mm3
* Hemoglobin level> 10g / 100ml
* Platelets> 50,000 / μl
* Weight> 40Kg
* Informed and signed consent;
* Patient affiliated to a social security scheme

Exclusion Criteria:

For liver transplant patients:

- Hepatocellular carcinoma or history of another cancer;

For kidney transplant patients:

- Kidney cancer or a history of another cancer

Common criteria:

* Active infectious diseases: positive serology for hepatitis A, B or C, HIV, HTLV, CMV and EBV;
* Associated autoimmune disease, including type 1 diabetes;
* GB <1500 / mm3;
* Any contraindication to citrate and calcium gluconate.
* Pregnancy or lactating woman
* Patient under guardianship or curatorship
* Patient deprived of liberty or under administrative security measure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Validate 4 preclinical batches of Treg cells from 2 liver transplant patients and 2 kidney transplant patients | At day 10
  Treg cells produced according to the expansion protocol defined by verifying the compliance of the batches according to the requirements of the guidelines on Good Manufacturing Practice specific to Advanced Therapy Medicinal Product) by respecting the validation and batch release criteria defined in this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: MIYARA Makoto, MD, PhD, Principal Investigator — AP-HP - Pitié Salpêtrière hospital
Locations (1):
- Pitié Salpêtrière hospital, Paris, France